CLINICAL TRIAL: NCT02495454
Title: GA101-miniCHOP Regimen for the Treatment of Elderly Unfit Patients With Diffuse Large B-cell Non-Hodgkin's Lymphoma A Phase II Study of the Fondazione Italiana Linfomi (FIL)
Brief Title: GA101-miniCHOP Regimen for the Treatment of Elderly Unfit Patients With Diffuse Large B-cell Non-Hodgkin's Lymphoma
Acronym: FIL_GAEL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary objective not obtained after interim analysis
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_GAEL; 2014-005697-10 (EudraCT Number)
Record Dates: First submitted 2015-06-08; First posted 2015-07-13 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-08

CONDITIONS: CD20 Positive Diffuse Large B-cell Lymphoma; Elderly Unfit Patients
MeSH Terms: interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ga101-miniCHOP (Experimental): 6 courses of GA101-miniCHOP regimen and 2 additional infusions of GA101, every 21 days (for a total of 6 courses of miniCHOP and 10 infusions of GA101).
  GA101-miniCHOP regimen:
  * Cycle 1 GA101: 1000 mg day 1, day 8 and day 15, iv Cyclophosphamide: 400 mg/mq, day 1, iv Doxorubicin: 25 mg/mq, day 1, iv Vincristine: 1 mg, day 1, iv Prednisone: 40 mg/mq, days 1-5, os
  * Cycles 2-6 GA101: 1000 mg day 1, iv Cyclophosphamide: 400 mg/mq, day 1, iv Doxorubicin: 25 mg/mq, day 1, iv Vincristine: 1 mg, day 1, iv Prednisone: 40 mg/mq, days 1-5, os
  * Two additional infusions of GA101: 1000 mg day 1, iv, every 21 days.
  Interventions: Drug: Ga101

INTERVENTIONS:
Drug: Ga101
  Other Names: Obinutuzumab

SUMMARY:
GA101-miniCHOP regimen for the treatment of elderly unfit patients with diffuse large B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Considering that the treatment of elderly unfit patients with DLBCL cannot be based on a full course of R-CHOP (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone), and that using a less intense R-miniCHOP (an attenuated version of the standard R-CHOP: Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone) combination an acceptable cure rate can be achieved this study is designed to try to improve the cure rate in unfit patients with DLBCL (Diffuse Large B Cell Lymphoma) by adopting the R-miniCHOP scheme substituting Rituximab with the more active GA101 monoclonal antibody. The study hypothesis is that a higher activity of the treatment can be achieved without modifying the cytotoxic part of the treatment but using a more active immunotherapy. Differently from the previous experience with R-miniCHOP eligible patient are not only identified using anagraphic criteria but adopting CGA (Comprehensive Geriatric Assessment) as part of initial assessment and considering as eligible unfit patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven CD20 positive Diffuse Large B-cell Lymphoma and Follicular grade III B lymphoma, according to WHO (World Health Organization) classification (local pathologist)
2. Age ≥ 65 years
3. No previous treatment
4. CGA assessment (Comprehensive Geriatric Assessment) performed before starting treatment
5. Unfit patients defined as follows:

   Age > 80 years with Fit profile, i.e. ADL (Activity of Daily Living) =6 residual functions IADL (Instrumental Activity of Daily Living) =8 residual functions CIRS (Cumulative Illness Rating Scale): no comorbidity of grade 3-4 and <5 of grade 2 or Age < 80 with Unfit profile, i.e ADL(Activity of Daily Living) > 5 residual functions IADL (Instrumental Activity of Daily Living) > 6 residual functions CIRS (Cumulative Illness Rating Scale): no comorbidity of grade 3-4 and 5-8 co-morbidities of grade 2
6. Ann Arbor Stage I with bulky, II-IV
7. At least one bi-dimensionally measurable lesion defined as > 1.5 cm in its largest dimension on CT scan
8. ECOG (Eastern Cooperative Oncology Group) performance status of 0, 1, or 2
9. Adequate hematologic function (unless caused by bone marrow infiltrate), defined as follows:

   Hemoglobin ≥ 10 g/dL Absolute neutrophil count ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L
10. LVEF (Left Ventricular Ejection Fraction) >50%
11. Ability and willingness to comply with the study protocol procedure
12. Life expectancy > 6 months
13. Accessibility of patient for treatment and follow up
14. Written informed consent

Exclusion Criteria:

1. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
2. Contraindication to any of the individual components of CHOP (Cyclophosphamide, Doxorubicin, Vincristine, Prednisone), including prior receipt of anthracyclines
3. History of other malignancies within 5 years prior to study entry except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer
4. Stage I without bulky
5. Patients with transformed lymphoma
6. Prior therapy for DLBCL (Diffuse Large B Cell Lymphoma), with the exception of nodal biopsy or local irradiation
7. Previous exposure to cytotoxic agents
8. Suspect or clinical evidence of CNS (Central Nervous System) involvement by lymphoma
9. HBsAg (Hepatitis B surface antigen), HCV (Hepatitis C Virus) or HIV (Human Immunodeficiency Virus) positivity; isolated HBcAb (Hepatitis B surface antibody) positivity is accepted only with concomitant treatment with Lamivudine
10. AST /ALT (Aspartate Aminotransferase/Alanine Aminotransferase)> twice upper the normal range; bilirubin > twice upper the normal range; serum creatinine > 2.5 mg /dl (unless these abnormalities were related to the lymphoma)
11. Evidence of any severe active acute or chronic infection
12. Concurrent co-morbid medical condition which might exclude administration of full dose chemotherapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Merli, MD, Principal Investigator — Ematologia - IRCCS Arcispedale Santa Maria Nuova
Locations (16):
- Italy (16):
  - A.O. Spedali Civili, Brescia, BS
  - AUSL di Ravenna, Ravenna, RA
  - Asmn-Irccs, Reggio Emilia, RE
  - Ematologia 1U - AO Città della Salute e della Scienza, Torino, TO
  - A.O. S. Maria di Terni, Terni, TR
  - A.O. SS. Antonio e Biagio e C. Arrigo, Alessandria
  - A.O. Universitaria Ospedali Riuniti - Ospedale Umberto I Di Ancona, Ancona
  - A.O. Ospedale Degli Infermi, Biella
  - Area Vasta Romagna e IRST, Meldola (FC)
  - IRCCS, Istituto Nazionale dei Tumori, Milan
  - A.O. Universitaria Policlinico Di Modena, Modena
  - SCDU Ematologia - Università del Piemonte Orientale, Novara
  - Irccs Istituto Oncologico Veneto (Iov), Padua
  - Oncoematologia e TMO Dopartimento Oncologia La Maddalena, Palermo
  - Ausl Di Rimini, Rimini
  - Ematologia - OSPEDALE DI CIRCOLO E FONDAZIONE MACCHI, Varese

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One case excluded for violation of inclusion criteria (transformed lymphoma)
Groups:
- Single Arm: 6 courses of GA101-miniCHOP regimen and 2 additional infusions of GA101, every 21 days (for a total of 6 courses of miniCHOP and 10 infusions of GA101) miniCHOP: an attenuated version of the standard CHOP, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone
Period: Overall Study
Arm/Group | Single Arm
Started | 34
Completed | 33 (One case excluded for violation of inclusion criteria (transformed lymphoma))
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: 6 courses of GA101-miniCHOP regimen and 2 additional infusions of GA101, every 21 days (for a total of 6 courses of miniCHOP and 10 infusions of GA101)
Arm/Group | Single Arm
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 33
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 82 [79 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 33
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 12.9 [11.0 to 13.5]
Stage [Count of Participants; unit: Participants] — Ann Arbor Staging:
  Stage I: nvolvement of a single lymph node region or lymphoid structure. Stage II: Involvement of two or more lymph node regions on the same side of the diaphragm.
  Stage III: Involvement of lymph regions or structures on both sides of the diaphragm.
  Stage IV: Involvement of extranodal site(s) beyond that designated as an involvement of a single, extranodal site contiguous or proximal to known nodal site.
  Bone marrow or liver involvement will always be considered as stage IV.
  Participants
    II | 6
    III | 11
    IV | 16
Bone Marrow Involvement [Count of Participants; unit: Participants]
  Negative | 27
  Positive | 6
Symptoms [Count of Participants; unit: Participants] — The presence of (a) unexplained weight loss of more than 10% of the body weight during the 6 months before initial staging investigation and/or (b) unexplained, persistent, or recurrent fever with temperatures above 38 C during the previous month and/or (c) recurrent drenching night sweats during the previous months is denoted by the suffix letter 'B'. 'A' indicates the absence of these symptoms
  Participants
    Absence of symptoms | 27
    Presence of symptoms | 6
ECOG PS (Eastern Cooperative Oncology Group Performance Status) [Count of Participants; unit: Participants] — ECOG Performance Status grade:
  0 Able to carry out all normal activity without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out light work
  2. Ambulatory and capable of all self-care but unable to carry out any work; up and about more than50% of waking hours
  3. Capable of only limited self-care; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair
  Participants
    0 | 12
    1 | 19
    2-3 | 2
LDH (lactate dehydrogenase) [Count of Participants; unit: Participants] — Ratio between measured level of LDH with the upper limit of normality. LDH levles with ratio <=1 was considered normal, LDH levels with ratio >1 was considered elevated.
  Participants
    <= Upper Limit | 10
    > Upper Limit | 23
International Prognostic Index [Count of Participants; unit: Participants] — International Prognostic Index (IPI): ranging fron 0 to 5. In this study was grouped 0-1 Low risk, 2 Intermediate risk, 3/5 High risk.
  Participants
    0-1 | 4
    2 | 8
    3/5 | 21
Comprehensive Geriatric Assessment [Count of Participants; unit: Participants] — Comprehensive Geriatric Assessment (CGA):
  FIT patients, without any co-morbidity; UNFIT patients, with mild co-morbidities; FRAIL patients, with severe co-morbidities.
  Participants
    UNFIT | 28
    FRAIL | 5

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CRR). Based a Central Independent Review Committee Considering Use the Conventional CT Scan Images.
Description: Complete Response Rate after 10 infusions of GA101 and 6 cycles of miniCHOP. Complete Remission (CR): Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, normalization of biochemistry abnormalities. If the bone marrow was involved by lymphoma before treatment, the infiltrate must be cleared on repeat bone marrow aspirate and biopsy of the same site. Partial disease (PR): >= 50% decrease in node diameter of the six largest dominant nodes or nodal masses and no new sites of disease; Stable disease (SD): is defined as less than a PR but is not progressive disease. Progession disease (PD): >50% increase diameter of node from nadir of any previously identified abnormal node nonresponders, and/or appearance of any new lesion.
Time Frame: Up to 36 months.
Population: Patients who received at last 1 cycle of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 33
Participants
  Complete Response | 14
  Partial Response | 8
  Stable Disease | 2
  Progression Disease | 8
  Not Assessed | 1

2. Secondary Outcome: Adverse Events (AEs)
Description: Rate of Adverse Events. Although was not defined a formal threshold, in this section we reported the summary of frequencies of maximum CTCAE observed in patients. Each patient was counted only once within the AE terms during the therapy. If, during the therapy the patient experiences more than one AE, only the AE with the greatest intensity was included in the summary.
Time Frame: Up to 36 months
Population: Patients who received at least 1 cycle of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 33
Participants
  CTCAE Grade 0 | 5
  CTCAE grade 1-2 | 11
  CTCAE grade >2 | 17

3. Secondary Outcome: Partial Response Rate (PRR)
Description: Partial Response Rate (PRR): patients in Partial Response after induction therapy.
  Frequency of PRR already reported in the table of principal end-point.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 33
Participants
  Partial Remission | 8
  Not in partial remission | 25

4. Secondary Outcome: ORR (Overall Response Rate)
Description: ORR (Overall Response Rate): sum of patiens with Complete or Partial response after the induction therapy.
Time Frame: Up to 36 months
Population: Patients who received at leat 1 cycle of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 33
Participants
  ORR | 22
  Less than ORR | 11

5. Secondary Outcome: OS (Overall Survival)
Description: OS (Overall Survival): defined as the time from the date of treatment start into the study until the date of death irrespective of cause. Patients who have not died at the time of end of the whole study, and patients who are lost to follow up, will be censored at the date of the last contact.
Time Frame: Up to 36 months
Measure: Mean (95% Confidence Interval); unit: Probability at 24 months
Arm/Group | Single Arm
Number analyzed (Participants) | 33
Probability at 24 months | 0.69 [0.50 to 0.82]

6. Secondary Outcome: PFS (Progression Free Survival)
Description: PFS (Progression Free Survival): defined as the time from entry into the study until lymphoma relapse/ progression or death as a result of any cause. Responding patients, patients who are lost to follow up, who withdrawal the consent or drop-out due to adverse event will be censored at their last assessment date. Patients died due to tumor will be considered in progression. Patients died for any other cause will be censored to the death date.
Time Frame: Up to 36 months
Measure: Mean (95% Confidence Interval); unit: Probability at 24 months
Arm/Group | Single Arm
Number analyzed (Participants) | 33
Probability at 24 months | 0.53 [0.34 to 0.68]

7. Secondary Outcome: Activities of Daily Living (ADL)
Description: Change in Activities of daily living score. The score ranging from 0 (bad performance) to 6 (good performance)
Time Frame: Up to 36 months
Reporting Status: Not Posted

8. Secondary Outcome: Instrumental Activities of Daily Living (IADL)
Description: Change in Instrumental Activities of Daily Living score. The score ranging from 0 (bad performance) to 8 (good performance).
Time Frame: Up to 36 months
Reporting Status: Not Posted

9. Secondary Outcome: Cumulative Illness Rating Scale (CIRS)
Description: Change in Cumulative Illness Rating Scale. The grading of comorbidity ranging from 0 (absent) to 4 (severe).
Time Frame: Up to 36 months
Reporting Status: Not Posted

10. Secondary Outcome: Questionnaire for Quality of Life (EORTC QLQ C30)
Description: Change in quality of life (QoL)
Time Frame: Up to 36 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 50 months
Groups:
- Single Arm: 6 courses of GA101-miniCHOP regimen and 2 additional infusions of GA101, every 21 days (for a total of 6 courses of miniCHOP and 10 infusions of GA101).
  NOTE: One SAE (atrial fibrillation) was recorded in patient excluded from analysis (not eligible for transformed lymphoma), exit before starting the 1st cycle of treatment.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 11/33
Serious Adverse Events (participants affected / at risk) | 6/33
Other Adverse Events (participants affected / at risk) | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=33)
Femur fracture (General disorders) | 2 (6)
Nausea (Gastrointestinal disorders) | 1 (6)
Congestive heart failure (Cardiac disorders) | 2 (6)
-sepsis (Infections and infestations) | 4 (6)
BCPO-Heart failure (Cardiac disorders) | 1 (6)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (6)
Non small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (6)
Lumbar pain, vertebral collapse (Musculoskeletal and connective tissue disorders) | 1 (6)
Atrial fibrillation (Cardiac disorders) | 1 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=33)
Anemia (Blood and lymphatic system disorders) | 6 (30)
Leukopenia (Blood and lymphatic system disorders) | 4 (30)
Neutropenia (Blood and lymphatic system disorders) | 15 (30)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (30)
Cardiac disorders (Cardiac disorders) | 5 (30)
Gastrointestinal disorders (Gastrointestinal disorders) | 12 (30)
General disorders (General disorders) | 6 (30)
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (30)
Infections (Infections and infestations) | 7 (30)
Injury (Injury, poisoning and procedural complications) | 2 (30)
Investigations (Investigations) | 3 (30)
Metabolism (Metabolism and nutrition disorders) | 8 (30)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (30)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (30)
Nervous system (Nervous system disorders) | 7 (30)
Renal (Renal and urinary disorders) | 2 (30)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 5 (30)
Vascular (Vascular disorders) | 1 (30)
Other (General disorders) | 8 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor, in accordance with art.5 of DM, minist. decree (Feb8,2013), guarantees the publication of the results of the study without any constraints and ensuring all the participating centres a proportional visibility to the actual participation. The single centre will be able to publish partial data of patients treated at the centre after the publication of the global results, or 24 months after the last patient's enrolment date, regardless of which centre the last patient was recruited at.

DOCUMENTS (2):
  • Study Protocol (2014-09-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT02495454/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/54/NCT02495454/SAP_001.pdf